CLINICAL TRIAL: NCT05805241
Title: Pharmacogenetics Analysis in Newborn Patients on Mechanical Ventilation and Fentanyl Administration
Brief Title: Pharmacogenetics Analysis of Fentanyl Administered in Newborns
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 31/22
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Fentanyl; Newborn; Pharmacogenetics
Keywords: Fentanyl; Newborn; Pharmacogenetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1 cc of blood sample, EDTA tube for:
  * DNA extraction with Qiagen Symphony kit
  * Genotyping using Illumina Omni 2.5 + exome array
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fentanyl is an opioid drug used as analgesic and anaesthetic also in Neonatal Intensive Care Units (NICU), according to the last national and international recommendations, during invasive life support strategies such as mechanical ventilation. Opioids manifest their sedative effect through activation of μ-opioid receptors, which are abundant both in the central and peripheral nervous system. Comparing fentanyl to morphine we can appreciate a much more powerful effect (75-220 major) with lower doses to obtain similar analgesic effect; these characteristics are due to the high lipophilicity of the molecule which easily crosses the blood-brain barrier (BBB). At the same time, fentanyl shows less adverse effects than morphine such as vomiting, nausea, gastrointestinal constipation, respiratory depression, dependence and tolerance. The drug is extensively metabolized by liver enzymes.

In routinary clinical practice it has been observed that large interindividual differences are found in the daily dosages needed to achieve pain control. Literature evidences that pharmacodynamic variation related to genotypes in receptor signalling or pain modulators may play an important role in this variability. Many genes are related to fentanyl pharmacodynamics and pharmacokinetics. Some polymorphism in these genes are already known to correlate with toxicity or efficacy of the drug, also in the paediatric population. More polymorphisms could be involved in abnormal pharmacodynamic or pharmacokinetics of fentanyl, therefore studies are necessary to better explain the possible role of pharmacogenetics in precision medicine especially in a very specific population as newborn.

ELIGIBILITY:
Inclusion Criteria:

1. all newborns on mechanical ventilation receiving fentanyl
2. parental written informed consent for participation in the study must be obtained

Exclusion Criteria:

1. Concurrent or previous opioid and/or midazolam administration (72 h interval required)
2. Known genetic or chromosomal anomaly
3. Probable rapid extubation

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns admitted in NICU and mechanically ventilated (MV) who received fentanyl administration for procedural pain.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Identification of already described polymorphisms | Within 6 hours of fentanyl administration
  To identify candidate polymorphisms based on the literature explaining interindividual variability in the pharmacokinetics and pharmacodynamics of fentanyl. 1 cc of blood sample will be collected
Identification of new polymorphisms | Within 6 hours of fentanyl administration
  To identify new polymorphisms explaining interindividual variability in the pharmacokinetics and pharmacodynamics of fentanyl. 1 cc of blood sample will be collected.

SECONDARY OUTCOMES:
To evaluate the statistical association between the polymorphisms identified and fentanyl dosage (µg/kg/hour) | Through study completion, an average of 18 months
  Association study. The univariate statistical analysis will consider the dose of fentanyl (µg/kg/hour) as a continuous dependent variable, associating it with the candidate genotypes (independent variables) by means of t-tests. The association of fentanyl dose with genotypes will also be evaluated in a multivariate model, adjusted for relevant demographic and clinical covariates, using generalized linear models.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Travan, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy